



## INFORMED CONSENT FOR PARTICIPANTS IN THE VALIDATION PROCESS OF ASTHMA-RELATED PICTOGRAMS FROM THE SIMAP PROJECT, THROUGH A RANDOMIZED CLINICAL TRIAL v2.0

The purpose of this document is to invite you to participate in the study titled "SIMAP: System for the automatic association of medical instructions with pictograms to facilitate understanding and retention." To help you make an informed decision, we will explain the procedures involved in conducting the research, as well as what your collaboration would entail:

- 1. Where and when the research will take place: The mentioned research will be conducted in ERA rooms belonging to CESFAM in Hualpén, Talcahuano, Valparaíso, and San Antonio.
- 2. Relevance of the study and benefits: When we visit the doctor or are discharged from medical care, we are usually given a list of instructions to follow, such as medication use, when to return to the doctor or emergency room, whether or not we can engage in physical activity, and what diet to follow. These instructions are provided in a short amount of time and in clinical language, which exposes us, as patients, to a lot of information. Often, we don't have enough time to fully understand it, which can affect how we follow our treatment. This project aims to develop a technological tool called SIMAP, which will assist healthcare personnel in delivering medical instructions more effectively. Each instruction will be accompanied by an image to help us understand more quickly how to use our medications. SIMAP will help us, as patients, to better understand and remember the medical instructions, providing us with more tools to correctly apply them at home and improve our health by adhering to the treatment.
- 3. Objectives: The objective of this study is to create a technological tool to assist healthcare personnel in primary care centers, specifically in ERA rooms belonging to CESFAM in Hualpén, Talcahuano, San Antonio, and Valparaíso, in communicating with patients. This will be done through the effective delivery of information using pictograms, which are images that help increase immediate understanding, retention, and adherence to treatment instructions, such as dosage, schedules, and types of medications.
- 4. What your participation entails: We invite you to participate in a study that aims to assess the understanding of medical instructions related to your asthma diagnosis. At the beginning of your participation in this study, a survey will be conducted to evaluate your level of control over bronchial asthma, and an interview will be conducted to gather general clinical information. If you agree to participate in this study, once your medical

RE-ACREDITADO

RES. EX N° 8080

REGIÓN DE BIO BIO

RECA HUD ABR 2022





check-up is complete, you will be given instructions for managing and treating your bronchial asthma, along with an educational brochure containing relevant information about your condition. At 7, 30, and 60 days after you begin your participation in the study, you will be asked to complete a survey to assess the level of control of your bronchial asthma and participate in an interview regarding the treatment and care of your bronchial asthma.

- 5. Risks: Your participation is considered to have minimal risks, mainly related to potential doubts about your current treatment. If this occurs, you will be referred to an appropriate instance to resolve them, at no cost to you.
- 6. Costs and payments: Participation in this database does not imply any additional charges for you or your family, either now or in the future.
- 7. Voluntariness: Your participation is completely voluntary, and you have the right to decline participation or withdraw your consent at any time. If you choose not to participate, you will not lose any rights as a patient of this institution, and the quality of the medical care you deserve will not be affected. If you withdraw your consent and initially agreed to participate with your identification, your personal and medical data that identify you will not be used. Additionally, all information obtained for the purposes of potential research will be deleted.
- 8. Participant Rights: If you have any questions about this study, please ask the surveyors, who will answer and clarify your doubts. If you still have questions, contact Rosa Figueroa from the University of Concepción at +56 (41) 2204247, or the alternate director from the University of Valparaíso, Dr. Carla Taramasco, at +569 (32) 250-7000. You are free to agree to participate and may withdraw from the study at any time by informing the surveyor or the project director or alternate director. If you decide to withdraw from the study, there will be no negative consequences regarding your care, medical treatment, or your status as a patient at the healthcare center you attend.
- 9. Confidentiality of the participant's identity: Although the survey includes collecting your name, it will not be disclosed. For analysis and future studies, your name will be replaced by a numerical code known only to authorized individuals involved in the study, who are required to keep it confidential.
- 10. Confidentiality of data: The information obtained through the surveys will be kept confidential and will be physically and digitally safeguarded by the lead investigator at the University of Concepción and by the co-investigator at the University of Valparaíso for five years. The results obtained will be provided to the management of the CESFAM under study.

RE-ACREDITADO

\*\* RES. EX.N° 8086

\*\* REGIÓN DE BIO BIO

\*\* CAHUNA ABR 2022





- 11. Use and Publication of Findings: The information obtained will remain confidential. It is possible that the results from the analysis of this data may be presented in medical journals and conferences; however, your name will not be disclosed.
- 12. Questions: If you have any questions about this medical research, you can contact the lead (+56 investigators, Dr. Rosa **Figueroa Iturrieta** 41 2204247, Taramasco rosa.figueroa@biomedica.udec.cl), Dr. Carla (+569 32 250-7000, carla.taramasco@uv.cl), or your treating physician. If you have questions about your rights as a participant in a medical research study, you may contact the president of the Scientific Ethical Committee of the Talcahuano Health Service, Dr. Patricia Marcela Cortés Jofré, at +56 41 272 21 50, or by sending an email to etica.sst@redsalud.gob.cl.

## **DECLARATION OF CONSENT**

- The purpose of this project, the procedures, the risks, the benefits, and my rights have been explained to me, including the right to withdraw my consent at any time I deem appropriate.
- I sign this document freely and voluntarily, without being forced to do so.
- I am not waiving any rights I have as a patient of this institution.
- I authorize the lead investigator and their collaborators to access and use the data contained in my medical records, surveys, and questionnaires for this study.
- I wish for my data to be stored: Anonymously With my personal identification
- I authorize being contacted in the future: Yes

DA DTICIDA NIT

• At the time of signing, I am given a signed copy of this document:

| PARTICIPANT: |
|---------------|
| Name: |
| Date: |
| Signature: |
| INVESTIGATOR: |
| Namo |

REACREDITADA

RES. EX Nº 6006

SEREM DE SALUD

RECIÓN DE BIO BIO

AL CAHAPA ABR 2022





| Date: |
|------------------------------------|
| Signature: |
| CENTER DIRECTOR OR THEIR DESIGNEE: |
| Name: |
| Date: |
| Signature: |

RE-ACREDITADO

RES EX Nº 8066

REGIÓN DE BIO BIO

REGIÓN DE BIO BIO

ACA HUD ABR 2022





REACREDITADO HITÉ ATIGO CIENTÍFICO

A CAHU

1° 6086 SALUD BIO BIO 2-2 ABR 2022

## CONSENTIMIENTO INFORMADO PARA PARTICIPANTES DEL PROCESO DE VALIDACIÓN DE PICTOGRAMAS RELATIVOS A ASMA DEL PROYECTO SIMAP, MEDIANTE ENSAYO CLINICO ALEATORIZADO.

V2.0

El propósito del presente documento es invitarlo a participar en el estudio titulado "SIMAP Sistema de asociación automática de indicaciones médicas a pictogramas para facilitar su comprensión y retención.". Para que usted pueda tomar una decisión informada, le explicaremos cuáles serán los procedimientos involucrados en la ejecución de la investigación, así como en qué consistiría su colaboración:

- Dónde y cuándo se llevará a cabo la investigación: La investigación mencionada se realizará en salas ERA pertenecientes a CESFAM de Hualpén, Talcahuano, Valparaíso y San Antonio.
- 2. Relevancia del estudio y beneficios: Cuando asistimos al médico o nos entregan una alta médica, generalmente, nos entregan, un listado de indicaciones a seguir, como, por ejemplo: uso de medicamentos, cuando volver a consultar al médico o sala de emergencia, si podemos o no realizar actividad física, alimentación a seguir. Estas indicaciones se entregan en un tiempo breve y con un lenguaje clínico, lo que hace que como pacientes nos expongamos a mucha información y muchas veces no tengamos tiempo de comprenderla, lo cual puede afectar la forma en que realizamos nuestro tratamiento.

Este proyecto pretende desarrollar una herramienta tecnológica llamada SIMAP, que apoye al personal de salud para que nos puedan entregar de mejor forma las indicaciones médicas. Cada indicación se acompañará de una imagen que nos ayuda a comprender de forma más rápida como usar nuestros medicamentos. SIMAP nos ayudará como pacientes a comprender y recordar de mejor manera las indicaciones médicas entregándonos más herramientas para aplicarlas bien en casa y mejorar nuestro estado de salud adhiriendo al tratamiento.

 Objetivos: El objetivo de este estudio es generar una herramienta tecnológica que apoye al personal de salud de centros de atención primaria, en especial salas ERA pertenecientes a CESFAM de Hualpén, Talcahuaro, San Antonio y

Versión 2.0 abril 2022







Valparaíso, en la comunicación con el paciente, mediante la entrega efectiva de información a través de pictogramas, que son imágenes que permitan aumentar la comprensión inmediata, retención y adhesión a las indicaciones asociadas al tratamiento, tales como dosis, horarios y tipo de medicamentos

- 4. En qué consiste su participación
  - En esta oportunidad lo invitamos a participar de un estudio que consiste en comprobar la comprensión de las indicaciones médicas relacionadas con su diagnóstico de asma. Para ello al inicio de su participación en este estudio, se le aplicará una encuesta para evaluar su grado de control del asma bronquial y una entrevista para conocer información clínica general. Si usted acepta participar en este estudio, una vez que finalice su control médico, se le entregarán las indicaciones para el manejo y tratamiento de su asma bronquial junto con un folleto educativo con información relevante a su condición. A los 7, 30 y 60 días después de iniciada su participación en el estudio, se le pedirá responder una encuesta para conocer el grado de control de su asma bronquial y una entrevista relativa al tratamiento y cuidado de su asma bronquial.
- 5. Riesgos: Se estima que su participación tiene riesgos mínimos asociados a dudas respecto a su actual tratamiento, si eso ocurriera, será derivado a una instancia pertinente para resolverlas, sin costo alguno para usted.
- 6. Costos y pagos: La participación de esta base de datos no significa cobro adicional de ningún tipo para usted o su familia, ni ahora ni en el futuro.
- 7. Voluntariedad: Su participación es completamente voluntaria y usted tiene el derecho a no aceptar participar o a retirar su consentimiento en cualquier momento que lo desee. Si usted no desea participar, no pierde ningún derecho que le asiste como paciente de esta institución y no se verá afectada la calidad de la atención médica que merece. Si usted retira su consentimiento, y acepto su participación manteniendo su identificación, los datos personales y médicos que lo identifiquen no serán utilizados. Además, toda la información obtenida con el propósito de posibles investigaciones será eliminado.
- 8. Derechos del participante: Si usted tiene alguna consulta sobre este estudio, por favor consulte a los encuestadores quienes responderán y aclararán sus dudas. En caso de aún tener dudas contacte a la directora-del proyecto Dra. Rosa Figueroa de la Universidad de Concepción al fono +96(41)220 directora alterna de la Universidad de Valparaíso Dra/Carla fono

Versión 2.0 abril 2022







+569 (32) 250-7000. Usted es libre de aceptar participar, y puede retirarse del estudio cuando usted lo desee comunicándolo al encuestador o a la directora o directora alterna del proyecto. Si usted decide retirarse del estudio no tendrá ninguna consecuencia negativa con respecto a su atención o tratamiento médico o su calidad de paciente en el centro de atención al que asiste.

- 9. Reserva de la identidad del participante Aunque la encuesta contempla recolectar su nombre, éste no será revelado. Para análisis y estudios posteriores su nombre será sustituido por un código numérico que solo conocerán personas autorizadas del estudio, quienes deben mantenerlo en reserva.
- 10. Confidencialidad de los datos: La información obtenida a través de las encuestas será confidencial y serán resguardadas física y digitalmente por la investigadora responsable en dependencias de la Universidad de Concepción y la coinvestigadora en las dependencias de la Universidad de Valparaíso durante cinco años. Los resultados obtenidos serán entregados a la Dirección del CESFAM en estudio
- 11. Utilización y Publicación de los hallazgos: La información obtenida se mantendrá en forma confidencial. Es posible que los resultados obtenidos del análisis de estas bases de dato sean presentados en revistas y conferencias médicas, sin embargo, su nombre no será revelado.
- 12. Preguntas: Si tiene preguntas acerca de esta investigación médica puede contactar a los investigadores responsables a la Dra. Rosa Figueroa Iturrieta (+56 41 2204247, rosa.figueroa@biomedica.udec.cl), Dra. Carla Taramasco (+569 (32) 250-7000, carla.taramasco@uv.cl), y/o su médico tratante. Si tiene preguntas acerca de sus derechos como participante en una investigación médica, usted puede hacerlo contactando al presidente del Comité Ético científico del Servicio de Salud de Talcahuano, Dra. Patricia Marcela Cortés Jofré, al teléfono +56 41 272 21 50 o enviando un correo electrónico a etica.sst@redsalud.gob.cl.

SEREMI DE SALUD REGIÓN DE BIO BIO



Versión 2.0 abril 2022





## **DECLARACION DE CONSENTIMIENTO**

- Se me ha explicado el propósito este proyecto, los procedimientos, los riesgos, los beneficios y los derechos que me asisten, incluido el derecho a retirar mi autorización en el momento que estime conveniente.
- Firmo este documento en forma libre y voluntaria, sin ser forzado/forzada a hacerlo.
- No estoy renunciando a ningún derecho que me asista como paciente de esta institución.
- Yo autorizo al investigador responsable y sus colaboradores a acceder y usar los datos contenidos en mi ficha clínica, encuestas y cuestionarios, para este

| estudio. | |
|---|---|
| Deseo que mis datos se almacenen: | |
| En forma anónima | |
| Con mi identificación personal | |
| Autorizo a ser contactado/a en el futuro Si No | |
| <ul> <li>Al momento de la firma se me entrega una copia firmada de este<br/>documento</li> </ul> | |
| PARTICIPANTE | |
| Nombre: Firma: | |
| Fecha: | |
| INVESTIGADOR | |
| Nombre: Firma: | |
| Fecha | |
| DIRECTOR DEL CENTRO O SU DELEGADO | |
| Nombre: Firma: | ĺ |
| Fecha: | |